CLINICAL TRIAL: NCT02887209
Title: A Pragmatic Pilot Study of Cognitive Behavioural Therapy for Insomnia Among People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Tyler Tulloch, PhD Student, Clinical Psychology, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSS
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Insomnia; HIV
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT-I (Experimental): This is a single arm study in which all participants receive the intervention (cognitive behavioural therapy for insomnia)
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — Cognitive behavioural therapy for insomnia (CBT-I; Edinger & Carney, 2008) is a standard 4-session cognitive behavioural therapy for insomnia administered biweekly in individual format. The first session involves presenting treatment rationale and introducing a behavioural treatment regimen consisting of a series of sleep habit parameters to follow, and determining a personalized "time in bed" prescription. The second session involves reviewing past-week sleep diary, discussing the role of cognitions in insomnia, and discussing constructive worrying techniques and the use of thought records. The third and fourth sessions are used to assist in adjusting "time in bed" prescriptions, to positively reinforce efforts, and to help problem-solve any problems they might have encountered.

SUMMARY:
Insomnia is a problem for approximately 75% of people living with HIV, which is much higher than the 6% to 10% of people with insomnia in the general population. It is currently unknown why the rate of insomnia is so high among people living with HIV, and because of this, they are often excluded from clinical trials examining the usefulness of cognitive behavioural therapy for insomnia (CBT-I), which is recommended as the first-line treatment for insomnia. Insomnia is also associated with poorer immune functioning and lower medication adherence. The purpose of this study is to examine whether CBT-I is useful at reducing insomnia among people living with HIV, and to examine whether this counselling is safe to provide to this population. Other purposes are to explore whether reducing insomnia will lead to improved immune functioning and medication adherence, to collect feedback about people's experiences receiving CBT-I, to examine which psychological and behavioural factors are associated with insomnia severity among people living with HIV.

DETAILED DESCRIPTION:
The prevalence of insomnia in the general population ranges from 6% to 10% (American Psychiatric Association, 2013), whereas its estimated prevalence among people living with HIV (PWH) is 73% (Rubinstein & Selwyn, 1998). Cognitive, behavioural, physiological, and psychosocial explanations for this elevated prevalence have been proposed (Taibi, 2013), however, there is a lack of consensus in the literature. Sleep disturbance is associated with disrupted immune functioning at the cellular level (Taylor, Lichstein, & Durrence, 2003), as well as increased risk of contracting infectious diseases (Patel et al., 2012); therefore, insomnia may be particularly problematic for PWH. Cognitive behavioural therapy for insomnia (CBT-I; Edinger & Carney, 2008) is the first-line treatment for insomnia (Qaseem et al., 2016; Schutte-Rodin et al., 2008), and medium to large effect sizes have been reported (Okajima et al., 2011). CBT-I is effective at treating insomnia among individuals with comorbid medical disorders such as chronic pain (Jungquist et al., 2012), fibromyalgia (Martínez et al., 2014), and cancer (Garland et al., 2014). Surprisingly, no study to date has examined the efficacy of CBT-I among PWH. The current study will evaluate the safety, feasibility, acceptability, and effects of CBT-I among 20 PWH using a pragmatic pilot study design. An exit interview will be conducted to elicit participant feedback about the treatment and methods used. Additional cross-sectional analyses will examine predictors of insomnia symptom severity and other sleep-related outcomes among a larger sample (n = 60). This will be the first study to examine the impact of CBT-I among PWH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to understand and communicate in English
* capable of providing informed consent
* presence of insomnia based on screener questionnaire cutoff score ≥ 15 on the Insomnia Severity Index
* HIV-seropositive
* willing to provide HIV viral load and CD4 count from blood work within the past two months

Exclusion Criteria:

* active suicidal ideation
* psychotic symptoms
* unmanaged bipolar disorder
* presence of a severe alcohol or substance use disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria
* hypnotic dependence
* presence of any breathing-related sleep disorders (obstructive sleep apnea hypopnea, central sleep apnea, and sleep-related hypoventilation), or circadian rhythm sleep-wake disorders
* working shift work or frequent time zone travel over the course of the study
* contingent or inconsistent hypnotic use, or anticipated change in hypnotic medication dose over the course of the study
* receiving psychotherapy for insomnia or any other mental disorder over the course of the study
* presence of an AIDS-defining opportunistic infection and/or a CD4 count < 200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Insomnia symptom severity | Two weeks post-treatment
  Insomnia symptom severity is measured using the Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
CD4+ (cluster of differentiation 4) cell count | Within two months post-treatment
  Obtained via self-report based on blood test results in past 3 months
HIV viral load | Within two months post-treatment
  Obtained via self-report based on blood test results in past 3 months
Combined antiretroviral therapy (cART) medication adherence | Two weeks post-treatment
  Measured using the Self-Rating Scale Item (SRSI) and Simplified Medication Adherence Questionnaire (SMAQ)
Sleep efficiency | Two weeks post-treatment
  Sleep efficiency is the amount of time spent sleeping vs. awake in bed
Total wake time | Two weeks post-treatment
  Total wake time is the total time spent awake between getting into bed at night

OTHER OUTCOMES:
Health-related quality of life | Two weeks post-treatment
  Measured using the Medical Outcomes Study Short-Form Health Survey (SF-36)
Depression symptom severity | Two weeks post-treatment
  Measured using the Centre for Epidemiological Studies in Depression Scale-Revised (CESD-R) and Depression Anxiety Stress Scales (DASS-21)
Treatment acceptability | Immediately post-treatment (final therapy session)
  Measured using the Therapy Evaluation Questionnaire (TEQ)
Intervention safety | Two weeks post-treatment
  Measured via qualitative exit interview, and includes any unwanted or adverse events associated with the intervention
Dysfunctional beliefs about sleep | Two weeks post-treatment
  Measured using the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16)
Sleep effort | Two weeks post-treatment
  Measured using the Glasgow Sleep Effort Scale (GSES)
Self-efficacy for sleep | Two weeks post-treatment
  Measured using the Self-Efficacy for Sleep Scale (SE-S)
Pre-sleep arousal | Two weeks post-treatment
  Measured using the Pre-Sleep Arousal Scale (PSAS-13)
Fatigue | Two weeks post treatment
  Measured using the Fatigue Severity Scale (FSS)
Anxiety Symptom Severity | Two weeks post treatment
  Measured using the Depression Anxiety Stress Scales (DASS-21)
HIV-Related Fatigue | Two weeks post treatment
  Measured using the HIV-Related Fatigue Scale (HRFS)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Tulloch, MA, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Department of Psychology, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garland SN, Johnson JA, Savard J, Gehrman P, Perlis M, Carlson L, Campbell T. Sleeping well with cancer: a systematic review of cognitive behavioral therapy for insomnia in cancer patients. Neuropsychiatr Dis Treat. 2014 Jun 18;10:1113-24. doi: 10.2147/NDT.S47790. eCollection 2014. PMID 24971014
- [Background] Jungquist CR, Tra Y, Smith MT, Pigeon WR, Matteson-Rusby S, Xia Y, Perlis ML. The durability of cognitive behavioral therapy for insomnia in patients with chronic pain. Sleep Disord. 2012;2012:679648. doi: 10.1155/2012/679648. Epub 2012 Aug 9. PMID 23470897
- [Background] Martinez MP, Miro E, Sanchez AI, Diaz-Piedra C, Caliz R, Vlaeyen JW, Buela-Casal G. Cognitive-behavioral therapy for insomnia and sleep hygiene in fibromyalgia: a randomized controlled trial. J Behav Med. 2014 Aug;37(4):683-97. doi: 10.1007/s10865-013-9520-y. Epub 2013 Jun 7. PMID 23744045
- [Background] Patel SR, Malhotra A, Gao X, Hu FB, Neuman MI, Fawzi WW. A prospective study of sleep duration and pneumonia risk in women. Sleep. 2012 Jan 1;35(1):97-101. doi: 10.5665/sleep.1594. PMID 22215923
- [Background] Qaseem A, Kansagara D, Forciea MA, Cooke M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Management of Chronic Insomnia Disorder in Adults: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2):125-33. doi: 10.7326/M15-2175. Epub 2016 May 3. PMID 27136449
- [Background] Rubinstein ML, Selwyn PA. High prevalence of insomnia in an outpatient population with HIV infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Nov 1;19(3):260-5. doi: 10.1097/00042560-199811010-00008. PMID 9803968
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] Taibi DM. Sleep disturbances in persons living with HIV. J Assoc Nurses AIDS Care. 2013 Jan-Feb;24(1 Suppl):S72-85. doi: 10.1016/j.jana.2012.10.006. PMID 23290379
- [Background] Taylor DJ, Lichstein KL, Durrence HH. Insomnia as a health risk factor. Behav Sleep Med. 2003;1(4):227-47. doi: 10.1207/S15402010BSM0104_5. PMID 15600216
- [Background] Edinger JD, Carney, CE. Overcoming insomnia: A cognitive-behavioral therapy approach. Therapist Guide. New York: Oxford University Press, 2008.
- [Background] Okajima I, Komada Y, Inoue Y. A meta-analysis on the treatment effectiveness of cognitive behavioral therapy for primary insomnia. Sleep and Biological Rhythms 9(1): 24-34, 2011.
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Washington, DC: Author.
- See also: Lab website — http://hivprevlab.ca